CLINICAL TRIAL: NCT06130865
Title: Responsiveness of Multiple Balance Assessment Tools in Patients With Peripheral Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/0246 Faria Ali Shahid
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Neuropathy
Keywords: Balance.; Diabetes; Diabetic Peripheral Neuropathy; Otago Exercise Plan
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Their is limited literature available regarding the assessment of balance by Fullerton Advanced Balance scale in patients with diabetic peripheral neuropathy, previous studies have only focused on the use of berg balance scale and mini-BESTest. So, this study aims to assess the responsiveness and sensitivity of Berg Balance Scale, Mini-BESTest, and Fullerton Advanced Balance Scale in the patients of diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetes is a serious, long-term condition with a major impact on the lives and well-being of individuals, families, and societies worldwide. Diabetic neuropathy is its most common clinical consequence. Diabetic Peripheral Neuropathy (DPN) is defined as "the presence of symptoms and/or signs of peripheral nerve dysfunction in people with diabetes after the exclusion of other causes." A person with DPN is up to 20 times more likely to fall than a non-diabetic of the same age, making falls an even more significant therapeutic concern. As a result of decreased balance, people with DPN are predisposed to falls, which can lead to injury, decreased balance confidence, fear-related avoidance of activities, and decreased quality of life. So, this study aims to assess the responsiveness and sensitivity of Berg Balance Scale, Mini-BESTest, and Fullerton Advanced Balance Scale in the population of DPN and it will also predict which of them is the most responsive and sensitive and first evaluates changes in balance of patients with DPN. After the comparison of responsiveness and sensitivity of these scales, it can predict the best tool for early assessment of balance impairment in the people with DPN. This study will be beneficial in early identification of fall risk and minimization of fall related injuries and complications.

ELIGIBILITY:
Inclusion Criteria:

* Either gender.
* Age between 40 to 60 years
* Known history of diabetes mellitus treated with by oral hypoglycemic drugs or insulin therapy.
* Known case of diabetic peripheral neuropathy (DPN)
* Patients who met the criteria of DN4 scored equal or greater than 4.
* Patients who have positive SHARPEND ROMBERG TEST.
* Balance impairment on BBS (21-40).

Exclusion Criteria:

* Lower limb muscles strength less than 3 on manual muscle testing.
* Any inflammatory condition, congenital or acquired malformation, vestibular system pathologies.
* Contraindication for engaging in physical activity (osteoarthritis, orthostatic hypo tension or any acute illness).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study Design:
  The study design is a prospective cohort study, where a group of participants will be followed over time to observe changes in patient outcomes after receiving physiotherapy interventions.
  Study Setting:
  Data for this study will be collected from the Irus Clinic and Rehabilitation Center Multan
  Study Duration:
  The study will span a period of six months, commencing after receiving approval from the Bioethical Review Board (BASR).
  Sample Size:
  The study will include a total of 104 participants.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 Weeks
  A clinical tool that assesses static and dynamic balance.
Mini Balance Evaluation Systems Test (mini-BESTest) | 8 weeks
  A clinical tool that assesses balance impairments by evaluating various components of balance control, including anticipatory postural adjustments, reactive postural responses, sensory orientation, and stability during gait.
Fullerton Advanced Balance Scale (FAB) | 8 weeks
  The FAB scale is a multi-item balance assessment test designed specifically to measure balance in higher-functioning active older adults.

CONTACTS AND LOCATIONS:
Overall Officials: aruba saeed, PHD, Principal Investigator — Riphah International University Pakistan
Locations (1):
- The Irus Clinic and Rehabilitation Center, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No